CLINICAL TRIAL: NCT03390062
Title: An One Arm, Open and Prospective Studyof Apatinib for the Treatment of Recurrent or Recurrent High-grade Glioma
Brief Title: A Study of Apatinib in Recurrent or Recurrent High-grade Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li ping, M.D., West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G-201702
Record Dates: First submitted 2017-12-19; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): apatinib 500 mg orally daily until the untolerabale toxicities、desease progress or death
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib, also known as YN968D1, is a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR2, also known as KDR). It is an orally bioavailable, small molecule agent which is thought to inhibit angiogenesis in cancer cells; specifically apatinib inhibits VEGF-mediated endothelial cell migration and proliferation thus blocking new blood vessel formation in tumor tissue.
  Other Names: Aitan

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of Apatinib for patients with Recurrent or Recurrent High-grade Glioma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, male or female;
* 2. The histologically confirmed first-line after the surgical resection of the WHOIII / IV glioma or previous surgery and / or radiotherapy and chemotherapy after the recurrence of WHOIII / IV glioma;
* 3. ECOG score: 0-2 points;
* 4. The main organs function properly, that is, meet the following criteria:(1) blood test:a. HGB≥90 g / L;b. ANC ≧ 1.5 × 109 / L;c. PLT ≥80 × 109 / L;(2) biochemical examination:a. ALB≥30g / L;b. ALT and AST <2*ULN;c. TBIL≤1.5*ULN; d. Plasma Cr≤1.5 *ULN;
* 5. No history of mental illness in patients;
* 6. Thyroid function is normal;
* 7. Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

* 1. Pregnant or lactating women;
* 2. Hypertensive patients who are not well controlled by antihypertensive medication (systolic blood pressure> 150 mmHg and diastolic blood pressure> 100 mmHg); those with grade I or greater myocardial ischemia or myocardial infarction, arrhythmia (including QT Period ≥ 440 ms) and grade I cardiac insufficiency, grading reference NCI-CTC AE 3.0;
* 3. Unable to swallow, chronic diarrhea and intestinal obstruction, significantly affect the medication and absorption;
* 4. Have a clear gastrointestinal bleeding concerns (such as local active ulcer lesions, fecal occult blood ++ above), within 6 months history of gastrointestinal bleeding;
* 5. Have mental illness, or history of substance abuse;
* 6. Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues; allowing the use of small doses of prophylaxis for prophylaxis, provided that the prothrombin time has an International Normalized Ratio (INR) ≤1.5 Farin (1 mg orally, once daily), low dose heparin (6,000 to 12,000 U daily for adults), or low dose aspirin (80 to 100 mg daily);
* 7. Researchers think it is not suitable for inclusion. All patients underwent CT or MRI of the head one week prior to the start of the protocol, with intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-04 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 24 month
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Progress-free Survival(PFS) | 24month
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 6month
  Proportion of patients with reduction in tumor burden of a predefined amount
EORTC QLQ-C30 | 24month
  The EORTC Quality of Life questionnaires are developed to assess the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: qing Mao, M.D., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided